CLINICAL TRIAL: NCT06442618
Title: Effectiveness of Extracorporeal Shockwave Therapy and Nutraceutical Supplementation in the Treatment of Epicondylitis: a Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Prof.ssa Giulia Letizia Mauro, Professor, University of Palermo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MFR042024
Record Dates: First submitted 2024-05-29; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-03

CONDITIONS: Epicondylitis, Lateral; Epicondylitis of the Elbow; Tennis Elbow
Keywords: Epicondylitis; Extracorporeal ShockWave Treatment (ESWT); Nutraceutical Supplementation; Rehabilitation; Musculoskeletal Disease; Tendinopathy; Tennis Elbow
MeSH Terms: conditions — Tennis Elbow; Musculoskeletal Diseases; Tendinopathy | interventions — Combined Modality Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Extracorporeal Shokwave Theraphy (Group A) (Active Comparator): Group A participants were invited to come to our department's outpatient clinics, wearing comfortable clothing. Meetings were held every six days, for a total of 5 sessions (30 days), lasting about 20 minutes each.
  Interventions: Other: Extracorporeal Shockwave Treatment (Group A)
- Nutraceutical Supplementation (Group B) (Active Comparator): Participants in Group B performed home therapy with nutraceutical supplementation containing: hyaluronic acid (200 mg), collagen (5,000 mg), manganese (10 mg) and vitamin C (250 mg), daily for 30 days; they were advised to always take it at the same time and independently of meals, so as not to interfere with absorption.
  Interventions: Other: Nutraceutical Supplementation (Group B)
- Combined Treatment (Group C) (Active Comparator): Participants in group C were invited to come to our department's outpatient clinics to perform treatment with focal ESWT; they had one session every six days for a total of 5 sessions lasting about 20 minutes each. Patients in this group took also additional nutraceutical therapy every day or 30 days.
  Interventions: Other: Combined Treatment (Group C)

INTERVENTIONS:
Other: Extracorporeal Shockwave Treatment (Group A) — Each session involved a 1:1 ratio of patient to physiatrist. The treatment modality was explained to the patient preliminarily, and before each session, the patients were clinically evaluated and the location of pain was identified.; so patients were asked to assume a comfortable position, and treatment with focal ESWTs was started as per the ISMST protocol
  Arms: Extracorporeal Shokwave Theraphy (Group A)
Other: Nutraceutical Supplementation (Group B) — Participants in Group B performed home therapy with nutraceutical supplementation containing: hyaluronic acid (200 mg), collagen (5,000 mg), manganese (10 mg) and vitamin C (250 mg), daily for 30 days. Patients were advised to shake the compound, before taking, and to store it at room temperature not exceeding 25 °C, in a cool, dry place, away from light and heat sources. The compound is also free of gluten and lactose, so it can be safely administered.
  Arms: Nutraceutical Supplementation (Group B)
Other: Combined Treatment (Group C) — Participants in group C were invited to come to our department's outpatient clinics to perform treatment with focal ESWT; they had one session every six days for a total of 5 sessions lasting about 20 minutes each. Patients in this group took also additional nutraceutical therapy; they took a daily supplemental treatment of hyaluronic acid, collagen, vitamin C and manganese for 30 days.
  Arms: Combined Treatment (Group C)

SUMMARY:
Lateral epicondylitis is a pathologic condition of the musculotendinous system, characterized by the presence of pain at the lateral epicondyle of the humerus; it is a tendinopathy of the extensor muscles of the forearm, often caused by overuse or repetitive use of the arm, forced extension of the elbow, or direct trauma to the humeral epicondyle. This study evaluated the efficacy of Extracorporeal ShockWave Treatment (ESWT) combined with a supplemental nutraceutical treatment of Hyaluronic Acid, Collagen, Vitamin C, and Manganese, compared with single treatment in patients with lateral epicondylitis in term of improvement in pain, functional capacity, muscle strength, and reduction of inflammation on ultrasound images. A clinical trial was conducted at the U.O.C. of "Recovery and Functional Rehabilitation" of A.O.U.P. "P. Giaccone" of Palermo from Marc 2024 to July 2024. Patients were randomized into 3 groups: in group "A", n° 5 sessions of focal ESWT were given every six days; in group "B", patients took daily for 30 days, supplemental nutraceutical treatment of Hyaluronic Acid, Collagen, Vitamin C, and Manganese; and group "C", patients had combined treatment of ESWT (one session every six days for a total of five sessions) and nutraceutical supplementation (one administration per day for one month). All patients were evaluated at enrollment (T0), after one month, at the end of rehabilitation treatment (T1), and at a follow up 30 days after the end of treatment (T2). Researched will compare patients treated with ESWT or with nutraceutical treatment, and patients who had combined treatment to see if there are real differences in term of pain reduction and improved short- and long-term quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of lateral epicondylitis;
* Ultrasound evidence of inflammatory status of the tendon of the wrist common extensor muscle;
* Numerical Rating Scale (NRS) at T0 ≥ 4;
* Pharmacological wash out starting seven days before treatment;
* Written informed consent.

Exclusion Criteria:

* Pregnancy;
* Already diagnosed or diagnostically defined neoplasms;
* Pacemaker wearers;
* Coagulation disorders and/or anticoagulant therapy;
* Skin lesions and/or local infections;
* Tendon injury and/or previous surgery on the wrist extensor tendons;
* Cervical myelopathy;
* Epilepsy;
* Patients with contraindications and/or allergies to the active ingredients of nutracetical supplementation;
* Obesity with BMI>30 (kg/m2).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Extent of pain: Numeric Rating Scale (NRS 0-10) | At the time of recruitment (T0) - After 30 day from the start of treatment (T1) - After 30 days from the end of treatment (T2)
  The NRS is a subjective scale that rates the extend of pain with a score between 0 and 10. a score of 10 corresponds to maximum pain.
Intensity of pain and disability: Patient-Rated Tennis Elbow Evaluation Scale (PRTEE) | At the time of recruitment (T0) - After 30 day from the start of treatment (T1) - After 30 days from the end of treatment (T2)
  This scale consists of 2 parts, namely pain (5 items) and functional activities (10 items). Each item has a score from 0 (no pain or difficulty in performing a task) to 10 (the worst pain or inability to perform a task). The total score is the combined score of the 2 parts

SECONDARY OUTCOMES:
Disability: Disability of the Arm, Shoulder and Hand (DASH) Questionnaire | At the time of recruitment (T0) - After 30 day from the start of treatment (T1) - After 30 days from the end of treatment (T2)
  This questinnaire is an important assessment tool, based on a district questionnaire, self-completed by the patient that aims to assess upper limb function; it consists of 38 questions, divided into 3 modules investigating different aspects of daily life, work activities, and sports/rehabilitation practices. The 38 items are scored from 1 to 5 (best score 1 and worst score 5) and refer to the patient's ability in the last 7 days
Handgrip strength | At the time of recruitment (T0) - After 30 day from the start of treatment (T1) - After 30 days from the end of treatment (T2)
  Handgrip strength was measured using a dynamometer; the patients squeezed the dynamometer maximally for 3 s. Three trials were attempted with 60 s of rest between each, and the average of all 3 grips were recorded.
Thickness of the common extensor tendon (CET) | At the time of recruitment (T0) - After 30 day from the start of treatment (T1) - After 30 days from the end of treatment (T2)
  The thickness of the common extensor tendon (CET) was assessed by ultrasound images.

CONTACTS AND LOCATIONS:
Locations (1):
- A.O.U.P. "P. Giaccone", Palermo, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Yang TH, Huang YC, Lau YC, Wang LY. Efficacy of Radial Extracorporeal Shock Wave Therapy on Lateral Epicondylosis, and Changes in the Common Extensor Tendon Stiffness with Pretherapy and Posttherapy in Real-Time Sonoelastography: A Randomized Controlled Study. Am J Phys Med Rehabil. 2017 Feb;96(2):93-100. doi: 10.1097/PHM.0000000000000547. PMID 27323324
- [Background] Pellegrino R, Di Iorio A, Filoni S, Mondardini P, Paolucci T, Sparvieri E, Tarantino D, Moretti A, Iolascon G. Radial or Focal Extracorporeal Shock Wave Therapy in Lateral Elbow Tendinopathy: A Real-Life Retrospective Study. Int J Environ Res Public Health. 2023 Feb 28;20(5):4371. doi: 10.3390/ijerph20054371. PMID 36901381
- [Background] Kinney WR, Anderson BR. Nonoperative Management of Lateral Epicondyle Tendinopathy: An Umbrella Review. J Chiropr Med. 2023 Sep;22(3):204-211. doi: 10.1016/j.jcm.2023.04.004. Epub 2023 Jul 10. PMID 37644995